CLINICAL TRIAL: NCT00630591
Title: DAMES: Daughters And MothErS Against Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00000466; 2007-0756 (Other: MD Anderson Cancer Center)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Daughters And MothErS Against Breast Cancer; DAMES; Breast Cancer; Weight Loss; Home-based weight loss; Quality of Life; Diet; Exercise; Daughter; Mother; Cancer Prevention; Prevention
MeSH Terms: conditions — Breast Neoplasms; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standardized Materials Group (Experimental)
  Interventions: Behavioral: Standardized Materials Group
- Independent Tailored Intervention (Experimental)
  Interventions: Behavioral: Independent Tailored Intervention
- Partner-Assisted Tailored Intervention (Experimental)
  Interventions: Behavioral: Partner-Assisted Tailored Intervention

INTERVENTIONS:
Behavioral: Standardized Materials Group — 7 sets of print materials will be mailed every 6-7 weeks. A short survey about the information received and how useful it was will be completed.
  Arms: Standardized Materials Group
Behavioral: Independent Tailored Intervention — Personalized notebooks and newsletters of diet and exercise information will be mailed. A short survey about the information received and how useful it was will be completed.
  Arms: Independent Tailored Intervention
Behavioral: Partner-Assisted Tailored Intervention — Daughters and Mothers, as a team, will each receive personalized notebooks and newsletters of diet and exercise information. A short survey about the information received and how useful it was will be completed.
  Arms: Partner-Assisted Tailored Intervention

SUMMARY:
Primary Aim:

-To explore the feasibility and acceptability of two distinctly different tailored, home-based diet and exercise interventions (one that relies on a partner-assisted, team-based approach that emphasizes the mother-daughter bond and one that is delivered to each independently) vs. standardized materials (attention control). This aim will be accomplished by assessing overall accrual, and by quantifying retention and adverse events in each study arm.

The study will be deemed feasible if it achieves the following criteria:

1. Accrual of 67 mother-daughter dyads into the intervention is accomplished within a 1-year period;
2. An attrition rate of less than 20% is achieved; and
3. The frequency of total adverse events is not significantly higher in either of the intervention arms (as compared to the attention control arm), and there is no more than one reported serious adverse event that is directly attributable to either of the interventions.

Detailed process data also will be collected on each intervention, i.e., use and perceived helpfulness of materials in promoting behavior change, frequency and quality of interaction between members of the mother-daughter dyad, feedback regarding intervention materials, etc.

Secondary Aim:

-To explore potential effects (and variation) noted among each of the three intervention arms from baseline to 6 and 12- month follow-up on the following endpoints: BMI, energy intake and nutrient density of the diet, exercise [min/week and metabolic equivalents (METs)], self-efficacy to adhere to an energy restricted, plant-based, low saturated fat diet and increased exercise, blood pressure, health-related quality of life (HRQOL), social support (in general and as specifically related to healthful dietary and exercise behavior), and characteristics of the mother-daughter bond (e.g., strength).

Secondary Aim:

-To explore potential mediators and moderators of healthful dietary and exercise behaviors, such as the strength of the mother-daughter bond, geographic proximity of mothers and daughters, self-efficacy for lifestyle change, etc.

DETAILED DESCRIPTION:
DAUGHTER AND MOTHER - FULL INTERVENTION STUDY:

Women who are overweight have a greater chance of developing breast cancer as they get older, and also are at greater risk of developing more aggressive cancer. Researchers want to study 3 different home-based diet and exercise weight loss programs and find out the effect of the programs on body weight, quality of life, and other health-related factors.

If you and your mother agree to participate in this year-long research study, you will be asked to sign this consent form and send it into our study office in the envelope provided. As soon as the study staff receives these forms from both you and your mother, they will contact you to schedule your first study visit.

First Study Visit:

If you live within 60 miles of the clinic, you will be asked to come in for an in-person appointment that lasts about 1 hour. During this visit, the study staff will measure your height, weight, blood pressure, and your waist (using a tape measure).

You will also be asked to have cardiopulmonary exercise testing, also known as a "stress test." The purpose of this test is to check your fitness level. During this test, you will pedal a stationary (exercise) bicycle. You will be asked to pedal at the same speed, as the difficulty is increased every minute. It will feel like you are pedaling up a hill that gets steeper and steeper. The test is stopped when you cannot pedal at the desired speed or you become too tired to pedal.

To accurately measure your fitness level, the study staff will measure the air that comes in and out of your mouth during exercise. You will be asked to wear a mouthpiece (similar to a snorkel used in deep sea diving) which is connected to a tube that sends the air you breathe out into a machine where it is tested. The exercise test will last about 8-12 minutes. As a safety precaution, during the test the study staff will also monitor your heart rate using a 12-lead electrocardiogram (ECG--a test that measures the electrical activity of the heart). This means that the study staff will place electrodes (sticky pads) at certain locations on your body so that they can monitor how your heart responds to exercise.

If you do not live within 60 miles of the clinic, or if you do not or cannot report to these medical centers, the study staff will send a study nurse to your house (or another location easy for you to reach) to measure your height, weight, blood pressure, and your waist (using a tape measure).

If the blood pressure measurement shows that your blood pressure is elevated (greater than 179/109), the study chair will need your personal doctor to say it is okay for you to take part in the study.

Activity Monitor and Phone Interviews:

After your first study visit, you will be given an activity monitor and instructions to wear it on your waistband or belt (like a pedometer), during the time you are awake, for 7 days in a row. The activity monitor will record your daily activity. At the end of the 7 days, you will be asked to return the activity monitor using a pre-addressed, postage-paid return envelope that you will be given to you with the monitor.

You will also receive a food poster and survey guide after your first study visit. You will use these to participate in 2 unscheduled telephone interviews within the next month. Each interview will take about 30 minutes. At the beginning of the interview, the interviewer will ask if the time is convenient for you, or if you need to reschedule the call for another time when you are available. During these interviews, you will be asked questions about your health and your diet and exercise behaviors.

Study Groups:

After both you and your mother have completed your surveys and the information from your activity monitor has been received by the study staff, both you and your mother will be randomly assigned as a team (like drawing names from a hat) to 1 of 3 intervention groups. All 3 interventions will not start sooner than 6 months after your mother's cancer diagnosis, to allow time for her to recover from treatment.

Standardized Materials Group:

If you are assigned to this group, you will be asked to exercise and to improve your diet to the best of your ability. In order to do this, you will receive 7 sets of print materials about diet, exercise, and other health information. These materials will be mailed every 6-7 weeks throughout the 1-year intervention period. After each mailing, you will be asked to complete a short survey (16 questions) about the information you received and how useful it was for you. You will be asked to return the survey in a prepaid, addressed envelope that was sent with the materials.

Independent Tailored Intervention Group If you are assigned to this group, you will be asked to exercise and to improve your diet to the best of your ability. In order to do this, you will receive a personalized notebook of diet and exercise information, which will be mailed to you at the start of the intervention. About every 6-7 weeks throughout the 1-year intervention period, you also will receive 6 personalized newsletters that will also provide you with more information. After each mailing, you will be asked to complete a short survey (16-20 questions) about the information you received and how useful it was for you. You will be asked to return the survey in a prepaid, addressed envelope that was sent with the materials.

In addition, you also will be given the following equipment and supplies to help you exercise and eat better:

* A pedometer, which is a small device worn just like the activity monitor that counts the number of steps you take each day;
* An Apple Nike + iPod® Sport kit (including iPod) that will play music to exercise to and record the time and distance you exercise;
* Food portion and fat information guides to help you make good food choices; and
* Logbooks that you will use to record what foods you eat and your exercise behaviors while you are on study.

Partner-Assisted Tailored Intervention Group:

If you are assigned to this group, you and your mother, as a team, will be asked to exercise and to improve your diets to the best of your ability. In order to do this, you will each receive a personalized notebook of diet and exercise information, which will be mailed to you at the start of the intervention. About every 6-7 weeks throughout the 1-year intervention period, you also will receive 6 personalized newsletters, which will also provide you and your mother with more information. After each mailing, you will be asked to complete a short survey (16-20 questions) about the information you received and how useful it was for you. You will be asked to return the survey in a prepaid, addressed envelope that was sent with the materials.

In addition, you and your mother also will be given the following equipment and supplies to help you exercise and eat better:

* A pedometer, which is a small device worn just like the activity monitor that counts the number of steps you take each day;
* An Apple Nike + iPod® Sport kit (including iPod) that will play music to exercise to and record the time and distance you exercise;
* Food portion and fat information guides to help you make good food choices; and
* Logbooks that you will use to record what foods you eat and your exercise behaviors while you are on study.

These materials that you will receive will emphasize a "team approach" to weight loss, and will encourage you and your mother to support one another. If you are assigned to this group, you will be encouraged to talk with your mother regularly. The study will reimburse you for up to 20 minutes/day of telephone calls between you and your mother. You will be told how to submit these phone charges if you are assigned to this group.

Follow-up Interviews and Visits:

At both 6 months and 1-year after you start this study, you will have a telephone interview with a member of the study staff. Each interview will last about 30 minutes, and will involve the same information collected during the 2 interviews at the beginning of study participation.

You will also be asked to take part in 2 more in-person visits (one at 6 months and another after a year) that will be like the visits performed at the beginning of the study.

Up to 134 women (67 mother-daughter pairs) will take part in this multicenter study. Up to 34 mother-daughter pairs will be enrolled at M. D. Anderson, and the rest will be enrolled at the Duke Comprehensive Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. DCIS or Stage I-IIIA Breast Cancer (MOTHERS)
2. Have a biological daughter at least 21 years old (MOTHERS)
3. Body Mass Index between 25 - 40 (MOTHERS) or 25 or above (DAUGHTERS)
4. English Speaking & Writing (MOTHERS & DAUGHTERS)
5. 5th grade or higher educational level (MOTHERS & DAUGHTERS)
6. Willingness to be randomized into the standardized or tailored intervention arms and to undergo baseline and follow-up assessments (MOTHERS & DAUGHTERS)
7. Must be at least 21 years of age (MOTHERS & DAUGHTERS)
8. Must reside within the United States, Puerto Rico or Guam and therefore able to participate in home visits made by Examination Management Services, Inc. (MOTHERS & DAUGHTERS)

Exclusion Criteria:

1. Evidence of progressive breast cancer or 2nd primaries (MOTHERS)
2. Pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program or to a diet high in fruits and vegetables, such as the following: untreated stage 3 hypertension; severe orthopedic conditions; scheduled for a hip or knee replacement within 6 months; paralysis; end-stage renal disease; dementia; unstable angina; heart attack, congestive heart failure or pulmonary conditions that have required hospitalization or oxygen within 6 months (MOTHERS & DAUGHTERS)
3. Currently exercising 30+ minutes/day for 5+ days/week (<150 minutes per week) (MOTHERS & DAUGHTERS)
4. Currently enrolled in a weight loss program (MOTHERS & DAUGHTERS)
5. Residing in institutionalized settings, e.g., living in assisted or skilled nursing facilities, and therefore not able to make independent choices about their lifestyle behaviors and participate fully in the intervention (MOTHERS AND DAUGHTERS).
6. Currently pregnant (MOTHERS & DAUGHTERS)
7. A previous diagnosis of breast cancer (DAUGHTERS).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Overall Accrual | 12-Months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - U.T. M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Demark-Wahnefried W, Jones LW, Snyder DC, Sloane RJ, Kimmick GG, Hughes DC, Badr HJ, Miller PE, Burke LE, Lipkus IM. Daughters and Mothers Against Breast Cancer (DAMES): main outcomes of a randomized controlled trial of weight loss in overweight mothers with breast cancer and their overweight daughters. Cancer. 2014 Aug 15;120(16):2522-34. doi: 10.1002/cncr.28761. Epub 2014 May 7. PMID 24804802
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org